CLINICAL TRIAL: NCT02917993
Title: An Open-Label Phase 1/2 Study of Itacitinib in Combination With Osimertinib in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: An Open-Label Phase 1/2 Study of Itacitinib in Combination With Osimertinib in Subjects With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-207; 2017-001750-34 (EudraCT Number)
Expanded Access: NCT05561985 (Available)
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; locally advanced; metastatic; epidermal growth factor receptor (EGFR) inhibition; Janus kinase inhibition
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Inhibition, Psychological | interventions — itacitinib; INCB039110; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Itacitinib + osimertinib (Experimental)
  Interventions: Drug: Itacitinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Itacitinib — In Phase 1, itacitinib at a protocol-defined starting dose, with subsequent dose escalation based on protocol-specific criteria. In Phase 2, itacitinib at the recommended dose from Phase 1.
  Other Names: INCB039110
Drug: Osimertinib — Osimertinib 80 mg once daily (QD)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of itacitinib in combination with osimertinib in subjects with locally advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at screening; outside the U.S. and European Union, an older limit could apply depending on local regulation (eg, 19 years and older for South Korea and 20 years and older for Taiwan).
* Histologically or cytologically confirmed unresectable locally advanced (Stage IIIB) or metastatic (Stage IV) NSCLC.
* Documented evidence of somatic activating mutation in EGFR (eg, G719X, exon 19 deletion, L858R, L861Q) in a tumor tissue sample. If a tissue sample is not available, then EGFR mutation status may be determined from circulating tumor DNA obtained from a blood sample using a validated or approved test kit.

  * Phase 1: Subjects must have previously received and progressed on or after treatment with an EGFR tyrosine kinase inhibitor (TKI). Additional lines of systemic therapy including investigational agents for locally advanced or metastatic NSCLC are allowed.
  * Phase 2: Subjects must not have received more than 1 prior line of therapy for locally advanced or metastatic NSCLC. First-line treatment must include an EGFR TKI, and subjects must have documented disease progression during or following treatment. Subjects with disease that progressed more than 6 months after completion of neoadjuvant/adjuvant chemotherapy or chemoradiation therapy are eligible if they received an EGFR TKI as first-line treatment for advanced NSCLC.

    * Subjects must have evidence of a T790M mutation in tumor tissue or plasma obtained after disease progression during or after treatment with an EGFR TKI. T790M mutation status from a local laboratory is acceptable; however, a tumor tissue sample or plasma sample suitable for centralized T790M mutation analysis must be available.
* Radiographically measurable or evaluable disease per RECIST v1.1.

Exclusion Criteria:

* Known CNS metastases, unless stable and asymptomatic. Subjects with CNS metastases may be eligible for the study, provided:

  * There is no evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases.
  * Subjects who are receiving corticosteroids must be on a stable or decreasing dose for at least 4 weeks before first dose of study treatment.
* Laboratory parameters outside the protocol-defined range.
* Clinically significant abnormalities found on an ECG.
* Clinically significant or uncontrolled cardiac disease.
* Past history of interstitial lung disease (ILD), drug induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
* Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive malignancy.
* Concurrent anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or hormonal therapy).
* Any previous use of Janus kinase (JAK) inhibitor, osimertinib, or other EGFR-directed therapy for T790M-mt NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Phase 1: Frequency, severity, and duration of adverse events (AEs) | From screening through 30-35 days after end of treatment, approximately 2 years.
Phase 1: Number of subjects with dose-limiting toxicities (DLTs) | Day 1 through Day 28
Phase 2: Objective response rate (ORR) based on RECIST v1.1 | Screening and 8-week intervals throughout the study, approximately 2 years.
  ORR defined as the percentage of subjects who have a confirmed best overall response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Maximum plasma concentration (Cmax) of itacitinib and osimertinib when administered in combination | Measured at protocol-defined study visits from Cycle 1 Day 1 through Cycle 1 Day 28.
Phase 1 and Phase 2: Area under the plasma concentration-time curve (AUC) of Itacitinib and osimertinib when administered in combination | Measured at protocol-defined study visits from Cycle 1 Day 1 through Cycle 1 Day 28.
Phase 2: Depth of response (DpR) based on RECIST v1.1 | Screening and 8-week intervals throughout the study, approximately 2 years.
  Defined as the percentage of maximal tumor shrinkage observed at the lowest point (nadir) compared with baseline.
Phase 2: Progression-free survival (PFS) | Interval from the first day of study treatment until disease progression or death due to any cause, approximately 3 years.
Phase 2: Overall survival (OS) | Interval from the first day of study treatment until death due to any cause, approximately 3 years.
Phase 2: Frequency, severity, and duration of AEs | From screening through 30-35 days after end of treatment, approximately 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, Study Director — Incyte Corporation
Locations (31):
- United States (23):
  - University of California San Diego, 3855 Health Sciences Drive, Mc 0987, La Jolla, California
  - University California San Francisco Thoracic Surgery and Oncology Clinic, 1600 Divisadero Street, Floor 4, San Francisco, California
  - Innovative Clinical Research Institute, 15111 Whittier Blvd., Suite 216, Whittier, California
  - Rocky Mountain Cancer Center, 1800 Williams Street, Suite 200, Denver, Colorado
  - Georgetown University Hospital, 3800 Reservoir Rd, NW, Washington D.C., District of Columbia
  - Lynn Cancer Center, 701 NW 13th Street, Floor 2, Boca Raton, Florida
  - Dana-Farber Cancer Institute, 450 Brookline Avenue, Boston, Massachusetts
  - Henry Ford Health System, 2799 W Grand Blvd., Detroit, Michigan
  - Karmanos Cancer Institute, 4100 John R. street mail Code HW04HO, Detroit, Michigan
  - Valley Hospital, 223 N Van Dien Avenue, Ridgewood, New Jersey
  - NYU Langone Medical Center, 160 East 34th Street, Floor 8, New York, New York
  - Stony Brook University Medical Center, 3 Edmund D. Pellegrino Road, Stony Brook, New York
  - Cleveland Clinic, 9500 Euclid Avenue, G Building, Cleveland, Ohio
  - Earle A. Chiles Research Institute Providence Cancer Center, 4805 NE Glisan Street, 2N35, Portland, Oregon
  - St. Luke's University Health Network, 701 Ostrum Street, Suite 403, Fountain Hill, Pennsylvania
  - Thomas Jefferson University, 111 S. 11th Street, Philadelphia, Pennsylvania
  - Texas Oncology - South Austin, 901 West 38th Street, Suite 200, Austin, Texas
  - University of Texas -MD Anderson Cancer Center, 1515 Holcombe Blvd., Houston, Texas
  - Texas Oncology - San Antonio Medical, 5206 Research Drive, San Antonio, Texas
  - Texas Oncology-Tyler, 910 E Houston Street, Suite 100, Tyler, Texas
  - Huntsman Cancer Institute, 2000 Circle of Hope Drive, Salt Lake City, Utah
  - US Oncology-Virginia Cancer Specialists, PC, 8503 Arlington Blvd., Suite 400, Fairfax, Virginia
  - West Virginia University Cancer Institute, 1 Medical Center Drive, Morgantown, West Virginia
- South Korea (3):
  - The catholic University of Korea, Seoul St. Mary's hospital, 222 Banpo-daero, Seoul, Seocho-gu
  - Severance Hospital, Yonsei University Health System 50-1 Yonsei-ro, Seoul, Seodaemun-gu
  - Asan Medical Center Department of Oncology, 88, Olympic-ro 43-gil, Seoul, Songpa-gu
- Spain (3):
  - Antiga Guarderia-Servei d'Oncologia Hospital Vall d'Hebron. P.Vall Hebron 119-129, Barcelona
  - Hospital Ramón y Cajal Ctra. Colmenar Viejo Km. 9,1 Planta (-)2 Dcha Oficina de Ensayos Clínicos Servicio de Oncología Médica, Madrid
  - Hospital Clinico Universitario Valencia Avenida Blasco Ibáñez 17 -8º, Valencia
- Taiwan (2):
  - Taipei Veterans General Hospital, No.201 Sec. 2 Shipai Rd l, Taipei, Beitou District
  - National Taiwan University Hospital, 7 Zhongshan South Road, Taipei, Zhongzheng District

REFERENCES:
- See also: An Open-Label Phase 1/ 2 Study of Itacitinib in Combination With Osimertinib in Subjects With Non-Small Cell Lung Cancer — https://incyteclinicaltrials.com/studies/incb-39110-207